CLINICAL TRIAL: NCT00683137
Title: Clinical Protocol for a Multiple Dose Randomized, Double-Blind, Placebo Controlled Study of the Analgesic Efficacy and Safety of Valdecoxib Compared to Placebo in Patients for Treatment of Post-Surgical Pain From Bunionectomy Surgery
Brief Title: Analgesic Efficacy And Safety of Valdecoxib For Treatment Of Post-Surgical Pain From Bunionectomy Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VALA-0513-144; A3471084
Record Dates: First submitted 2008-03-31; First posted 2008-05-23 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Pain; Hallux Valgus
MeSH Terms: conditions — Pain; Hallux Valgus | interventions — valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 3 (Active Comparator)
  Interventions: Drug: valdecoxib/placebo

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 40 mg tablet by mouth followed by a valdecoxib 20 mg tablet by mouth after 1 to 12 hours of the initial dose on Day 1 then a valdecoxib 20 mg tablet by mouth once daily on Days 2 through 5
  Arms: Arm 1
Drug: valdecoxib — valdecoxib 40 mg tablet by mouth followed by a valdecoxib 20 mg tablet by mouth after 1 to 12 hours of the initial dose on Day 1 then a valdecoxib 20 mg tablet by mouth twice daily on Days 2 through 5
  Arms: Arm 2
Drug: valdecoxib/placebo — valdecoxib 40 mg tablet by mouth followed by a valdecoxib 20 mg tablet by mouth after 1 to 12 hours of the initial dose on Day 1 then placebo on Days 2 through 5
  Arms: Arm 3

SUMMARY:
The study was done to evaluate the pain relief and safety of 2 valdecoxib doses compared to placebo in patients with moderate or severe pain following bunionectomy surgery, and to evaluate the effect of the 2 valdecoxib doses compared to placebo on health outcome measures and on the occurrence of opioid related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an uncomplicated primary unilateral first metatarsal bunionectomy surgery (with or without ipsilateral hammer toe repair) who required open manipulation of bone with periosteal evaluation under general anesthesia (Mayo block)
* Patients with a baseline pain intensity (VAS) of greater than or equal to 45 mm
* Patients with a baseline pain intensity (categorical) of moderate or severe

Exclusion Criteria:

* Patients scheduled to undergo other surgical procedures that would be expected to produce a greater degree of surgical trauma than the orthopedic procedure alone
* Treatment with patient-controlled analgesia (PCA) subsequent to the end of anesthesia
* Long-acting local anesthetics or local anesthetics coadministered with epinephrine injected into the index joint space
* Use of tricyclic antidepressants, tranquilizers, neuroleptics, neuroleptic antiemetics, COX-2 inhibitors, NSAIDs, and corticosteroids
* Use of NSAID or analgesia after midnight the night prior to surgery or unwilling to abstain from NSAIDs or other analgesics, except as specified in the protocol, during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2002-10; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Patient's Global Evaluation of Study Medication | Day 2 and Day 3
Summed Pain Intensity (SPI) (categorical) through 24 hours | Day 2 and Day 3

SECONDARY OUTCOMES:
Health Outcomes Post-Discharge Recovery Experience | Days 2 to 5
adverse events | continuous
Time to first dose of rescue medication (rescue analgesic medication) | Days 2 to 5
SPI 24 (categorical) | Day 4 and Day 5
Time-specific Pain Intensity (PI) (categorical) | Days 2 to 5
SPI 24 (Visual Analog Scale [VAS]) | Days 2 to 5
Time-specific PI (VAS) | Days 2 to 5
Patient's Global Evaluation of Study Medication | Day 4 and Day 5
Percent of patients who took rescue medication (rescue analgesic medication) | Days 2 to 5
Worst Pain Intensity (derived from the Modified BPI-Short Form) | Days 2 to 5
Time between doses of study medication | Days 2 to 5
Individual and Composite Pain Interference Score (derived from the modified BPI-Short Form) | Days 2 to 5
Symptom Distress Questionnaire | Days 2 to 5
Average Pain Intensity (derived from the Modified BPI-Short Form) | Days 2 to 5
Amount of rescue medication (rescue analgesic medication) taken | Days 2 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (53):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Milford, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Cooper City, Florida
  - Pfizer Investigational Site, Cutler Ridge, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Port Richey, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Spring Hill, Florida
  - Pfizer Investigational Site, Addison, Illinois
  - Pfizer Investigational Site, Elk Grove Village, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Annapolis, Maryland
  - Pfizer Investigational Site, Chester, Maryland
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Austintown, Ohio
  - Pfizer Investigational Site, Canfield, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Youngstown, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Havertown, Pennsylvania
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Reading, Pennsylvania
  - Pfizer Investigational Site, State College, Pennsylvania
  - Pfizer Investigational Site, Upland, Pennsylvania
  - Pfizer Investigational Site, Wyomissig, Pennsylvania
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Holladay, Utah
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Sandy City, Utah
  - Pfizer Investigational Site, St. George, Utah
  - Pfizer Investigational Site, Tacoma, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=VALA-0513-144&StudyName=Analgesic%20Efficacy%20And%20Safety%20of%20Valdecoxib%20For%20Treatment%20Of%20Post-Surgical%20Pain%20From%20Bunionectomy%20Surgery.%0A